CLINICAL TRIAL: NCT00074919
Title: Expanded Access Use of Myozyme (Alglucosidase Alfa) in Patients With Infantile-onset Pompe Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGLU02203
Record Dates: First submitted 2003-12-23; First posted 2003-12-25 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Glycogen Storage Disease Type II; Glycogenosis 2
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease; Acid Maltase Deficiency Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

INTERVENTIONS:
Biological: alglucosidase alfa — 20 mg/kg qow
  Other Names: Myozyme

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The objective of this protocol is to provide enzyme replacement therapy with rhGAA on an expanded access basis, to severely affected patients with infantile-onset Pompe disease for whom there is no alternative treatment and who do not meet the clinical characteristics described in the inclusion criteria for participation in other Genzyme Corporation-sponsored study currently enrolling patients with infantile-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient or the patient's legal guardian(s) must provide written informed consent prior to any study-related procedures being performed;
* The patient must have a diagnosis of infantile-onset Pompe disease as defined by: a) The patient has/had onset of symptoms compatible with Pompe disease by 12 months of age adjusted for gestation, if necessary. Age at onset of symptoms must be documented in the patient's medical record(s). AND b) The patient has documented GAA deficiency, i.e., below the laboratory-defined cut-off value as determined by the laboratory performing the GAA enzyme activity assay. Tissues used for determination of GAA deficiency may include blood, muscle or skin fibroblasts.
* Patients less than or equal to 6 months of age must have one of the following: a) Cardiomyopathy, defined as a LVMI determined by cross-sectional echocardiography; OR b) a requirement for invasive or non-invasive ventilatory support, where non-invasive ventilation is defined as any form of ventilatory support applied without the use of an endotracheal tube.
* Patients greater than 6 months of age must have 2 of the following: a) Cardiomyopathy, defined as a LVMI determined by cross-sectional echocardiography; b) a requirement for invasive or non-invasive ventilatory support, where non-invasive ventilation is defined as any form of ventilatory support applied without the use of an endotracheal tube; OR c) Severe motor delay, defined as failure to perform gross motor skills achieved by 90% of normal aged peers on the Denver Developmental Assessment;
* The patient or his/her legal guardian(s) must have the ability to comply with the clinical protocol.

Exclusion Criteria:

* Major congenital abnormality;
* Clinically significant organic disease (with the exception of symptoms relating to infantile-onset Pompe disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company

REFERENCES:
- [Derived] Kishnani PS, Goldenberg PC, DeArmey SL, Heller J, Benjamin D, Young S, Bali D, Smith SA, Li JS, Mandel H, Koeberl D, Rosenberg A, Chen YT. Cross-reactive immunologic material status affects treatment outcomes in Pompe disease infants. Mol Genet Metab. 2010 Jan;99(1):26-33. doi: 10.1016/j.ymgme.2009.08.003. PMID 19775921